CLINICAL TRIAL: NCT04287387
Title: Response of Gut Microbiota in Type 2 Diabetes to Hypoglycemic Agents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIMCAS2018001
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Type2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; gut microbiota; hypoglycemic drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Tablets; Acarbose; Sitagliptin Phosphate; dapagliflozin; Pioglitazone; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Glucophage group (Experimental)
  Interventions: Drug: Glucophage 500Mg Tablet
- Acarbose group (Experimental)
  Interventions: Drug: Acarbose Tablets
- Sitagliptin group (Experimental)
  Interventions: Drug: Sitagliptin tablet
- Dapagliflozin group (Experimental)
  Interventions: Drug: Dapagliflozin Tablet
- Pioglitazone group (Experimental)
  Interventions: Drug: Pioglitazone Tablets
- Glimepiride group (Experimental)
  Interventions: Drug: Glimepiride Tablets

INTERVENTIONS:
Drug: Glucophage 500Mg Tablet — 0.5g three times daily
  Arms: Glucophage group
Drug: Acarbose Tablets — 50mg three times daily
  Arms: Acarbose group
Drug: Sitagliptin tablet — 100mg once daily
  Arms: Sitagliptin group
Drug: Dapagliflozin Tablet — 10mg once daily
  Arms: Dapagliflozin group
Drug: Pioglitazone Tablets — 30mg once daily
  Arms: Pioglitazone group
Drug: Glimepiride Tablets — 2mg once daily
  Arms: Glimepiride group

SUMMARY:
Intestinal microflora refers to the trillions of microorganisms living in our gut, which is considered as an independent endocrine organ of human body. Intestinal microbiota plays a very important role in human health. The composition of human intestinal microbiota is affected by a variety of factors, including age, living region, eating habits, nutrition, probiotics, antibiotics and so on. It is found that the imbalance of intestinal microbiota is closely related to the occurrence and development of metabolic diseases including type 2 diabetes mellitus (T2DM). There are great differences in the structure and function of intestinal microbiota between healthy people and T2DM patients, and recently changes of intestinal microbiota have been observed in pre-diabetes. In recent years, it has been found that some commonly used hypoglycemic drugs may regulate and improve the imbalance of intestinal flora of T2DM patients, including metformin, α - glucosidase inhibitor, and Glucagon-like peptide-1(GLP-1) receptor agonist, which have a positive impact on the short chain fatty acid (SCFAs) producing bacteria. However, on the one hand, subjects of those studies were mostly western population and there were just a few studies on the influence of anti-diabetic drug on human gut microbiota in Chinese population, on the other hand, the study of influence of Dipeptidyl peptidase-4(DPP-4) inhibitors, sulfonylureas, sodium-dependent glucose transporters-2(SGLT-2) inhibitors or thiazolidinediones on intestinal microbiota is rare or even absent. This study aims to explore the effect of different hypoglycemic drugs on intestinal flora and find the potential intestinal target of drug action in Chinese population.

DETAILED DESCRIPTION:
In this study, T2DM patients who were free of anti-diabetic drugs or those have taken hypoglycemic drugs and ready to add a new drug were recruited, they were treated with metformin, α - glucosidase inhibitor, DPP-4 inhibitors, sulfonylureas, SGLT-2 inhibitors, or thiazolidinediones according to their state of illness. Faecal specimen will be collected for test of composition of gut microbiota at baseline and 4-week, 8-week，12-week after taking medication. At baseline, patients will take physical examination and blood test, every patient will complete the questionnaire under the direction of doctors to get their general information and diet habits. Physical examination and blood test will repeat at 4-week, 8-week，12-week after treatment.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of World Health Organization (WHO) in 1999, type 2 diabetes mellitus was diagnosed clinically
* The age ranged from 18 to 65 years (including 18 and 65 years)
* Free of hypoglycemic drugs in the past 3 months; or have taken hypoglycemic drugs, and other hypoglycemic drugs need to be added at present.
* Sign written consent form voluntarily

Exclusion Criteria:

* Other types of diabetes mellitus
* At least in the last 1 month, no antibiotics or microbial agents have been used
* History of infectious diseases such as tuberculosis, viral hepatitis, HIV, and periodontal disease; history of dental disease
* Acute complications of diabetes mellitus within 6 months
* History of myocardial infarction or stroke within 6 months, or existing severe cardiovascular disease and risk
* Abnormal liver function [i.e. serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 1.5 times higher than the upper limit of normal value]；Abnormal renal function [glomerular filtration rate≤60 ml/min]
* Severe hypertension that defined as systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥90 mmHg with drug therapy, or hypotension (resting seat blood pressure < 90/50 mmHg)
* History of acute and chronic gastroenteritis or gastrointestinal surgery
* psychosis, alcohol dependence or history of drug abuse, lactation women, participation in other studies three months before the trial, allergic constitution or allergic to a variety of drug and those researchers think inappropriate to the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-03-02 (Estimated); Primary Completion 2021-03-02 (Estimated); Study Completion 2021-03-02 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to post-treatment in composition in gut microbiota analyzed by meta-genome sequencing. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in fasting blood glucose. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in level of TNF-a. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in fasting insulin. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in blood lipid including cholesterol, triglycerides, high-density lipoprotein. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in 2-hour postprandial blood glucose. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in level of IL-6. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in level of IL-8. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in level of IL-10. | Baseline, Week 4, Week 8, Week 12
Changes from baseline to post-treatment in composition in level of C-reative protein. | Baseline, Week 4, Week 8, Week 12

SECONDARY OUTCOMES:
The linear relationship between gut microbiota and blood glucose and blood lipid level. | Week 4, Week 8, Week 12
The linear relationship between gut microbiota and inflammation factors level. | Week 4, Week 8, Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No